CLINICAL TRIAL: NCT04124523
Title: International Opinion Study on Peri-operative Cerebrospinal Fluid Leaks Management After Endoscopic Skull Base Surgery
Brief Title: Perioperative CSF Leak Management - an Opinion Study
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0468
Record Dates: First submitted 2019-10-03; First posted 2019-10-11 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2019-09

CONDITIONS: Cerebrospinal Fluid Leak
Keywords: skull base surger; CSF leaks; intracranial pressure; endoscopic skull base surgery; CSF depletion; ENT surgeon or neurosurgeon
MeSH Terms: conditions — Cerebrospinal Fluid Leak

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cerebrospinal fluid (CSF) leak is a rare condition. When it involves the ventral skull base, a surgical closure may be achieved using endoscopic skull base surgery techniques. The major principles remain in achieving a watertight closure that can also support the brain (and avoid brain sagging) in case of extensive skull base defects. Surgical techniques are well described. Many clinical factors may influence the successful rate of the reconstruction. However, there is a lack of clinical study on perioperative management of CSF leaks. The purpose of this study is to gather the opinion of skull base surgeons on the post-operative management of patients to avoid CSF leak recurrence.

•Methods: The investigators will collect data from skull base surgeons using an electronic survey questionnaire (Google Form, Google, Mountain View, California, U.S.A.) submitted by e-mail to the members of the French Association of Rhinology, to the European Rhinologic Society, to the French college of neurosurgeons, to the Italian skull base society members, and to the former students of the European endoscopic skull base diploma. This is an anonymous 60-items survey. Questions were classified in eight sections: general questions, material used at the end of the surgical procedure, post-operative resting position, drugs, CSF depletion, post-operative advices, explorations in case of early recurrence of the rhinorrhoea, and follow-up modalities.

•Discussion: The investigators aim to understand the actual practice of skull base surgeons after closure of ventral skull base CSF leaks. This can serve as a basis for conducting clinical studies in the future.

ELIGIBILITY:
Inclusion criteria

An individual must fulfill all of the following criteria in order to be eligible for study enrollment:

* Active skull base surgery practice (ENT surgeon or neurosurgeon)
* Volunteering

Non inclusion criteria

* Subject unable to read or/and write
* Undergraduate students
* Refusal to participate

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ENT surgeon or neurosurgeon skull base surgery practice
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of perioperative management of CSF leaks | 1 day (pre-treatment)
  Evaluation of perioperative management of CSF leaks at pre-treatment (preoperative) with 60 items questionnaire (QCM)
Evaluation of perioperative management of CSF leaks | 1 day (the end of the surgery)
  Evaluation of perioperative management of CSF leaks at the end of the surgery with 60 items questionnaire (QCM)
Evaluation of perioperative management of CSF leaks | maximum 2 weeks (during hospitalization)
  Evaluation of perioperative management of CSF leaks during hospitalization with 60 items questionnaire (QCM)

SECONDARY OUTCOMES:
Comparison of practices of surgeons according by specialties | 1 day (pre-treatment)
  Comparison of practices of surgeons according by specialties at pre-treatment (preoperative) with 60 items questionnaire (QCM)
Comparison of practices of surgeons according by specialties | 1 day (the end of the surgery)
  Comparison of practices of surgeons according by specialties at the end of the surgery with 60 items questionnaire (QCM)
Comparison of practices of surgeons according by specialties | maximum 2 weeks (during hospitalization)
  Comparison of practices of surgeons according by specialties during hospitalization with 60 items questionnaire (QCM)

CONTACTS AND LOCATIONS:
Overall Officials: Valentin Favier, MD, Principal Investigator — University Hospitals of Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC